CLINICAL TRIAL: NCT02687815
Title: Vitamin D to Prevent Severe Asthma Exacerbations
Brief Title: Vitamin D to Prevent Severe Asthma Exacerbations (Vit-D-Kids Asthma)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility of vitamin D supplementation based on protocol threshold: <30% conditional power to detect pre-specified effect- 16% reduction in severe exacerbations.
Sponsor: Juan Celedon, MD (Other)
Collaborators: Pharmavite LLC (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Juan Celedon, MD, Niels K. Jerne Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO12020541; U01HL119952 (NIH)
Record Dates: First submitted 2016-02-11; First posted 2016-02-22 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: Vitamin D, severe asthma exacerbations, children
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 (Experimental): Cholecalciferol (Vitamin D3) 4000 IU oral gel cap daily
  Interventions: Drug: vitamin D3 4000 IU
- placebo (Placebo Comparator): placebo formulations will be in gel cap form and identical to the active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vitamin D3 4000 IU — The vitamin D3 will be in oral gel cap form and contain 4000 International Units (IU) of cholecalciferol per gel cap.
  Other Names: Cholecalciferol
  Arms: vitamin D3
Drug: Placebo — The placebo is a gel cap that is indistinguishable from the vitamin D3 gel cap.
  Arms: placebo

SUMMARY:
This study will determine whether vitamin D3 prevents severe asthma attacks in children who have a serum vitamin D (25(OH)D) level <30 ng/ml and who are being treated with inhaled corticosteroids for asthma. Half the participants will receive vitamin D3 at a dose of 4,000 IU/day, and the other half will receive placebo.

DETAILED DESCRIPTION:
Results from experimental studies, observational studies, two small trials, and a recent meta-analysis suggest that vitamin D reduces the risk of severe asthma exacerbations, and that this protective effect may be due to immune modulation of viral illnesses and/or increased response to inhaled corticosteroids (ICS).

On the basis of those findings, the investigators hypothesize that vitamin D reduces the incidence of severe asthma exacerbations in high-risk school-aged children who have a serum vitamin D level <30 ng/ml and who are being treated with ICS for persistent asthma. The investigators further hypothesize that this protective effect results from reduced incidence of common viral illnesses or enhanced response to ICS. These hypotheses will be tested in a 48-week randomized double-masked placebo-controlled trial of vitamin D3 supplementation to prevent severe asthma exacerbations in 400 children aged 6 to 16 years who have vitamin D insufficiency or deficiency (a serum 25(OH)D <30 ng/ml) and experienced a severe exacerbation in the prior year (a marker of high risk for subsequent events), and who (after a run-in period) are well controlled on medium-dose inhaled corticosteroids.

Our primary aim will determine whether vitamin D3 (4,000 IU/day) reduces the risk of severe asthma exacerbations (our primary outcome) in participating children. Secondary aims will determine the efficacy of vitamin D3 supplementation in: 1) preventing severe asthma exacerbations due to viral infections, 2) reducing the daily and average cumulative dose of inhaled corticosteroids.

Study participation involves 8-9 visits, with each visit lasting between 30-90 minutes. Participation requires completion of study questionnaires, spirometry (breathing tests), and collection of blood samples (to measure vitamin D levels) and urine samples (to measure urinary calcium/creatinine ratios) at some study visits. Since the start of the study, vitamin D levels and urinary calcium/creatinine ratios have been simultaneously measured, to monitor for both vitamin D toxicity and high risk of severe vitamin D deficiency or rickets, which (should they occur) would be managed by a pediatric endocrinologist or a pediatric nephrologist, as appropriate.

All safety data for the study is regularly reviewed by a Data Safety Monitoring Board appointed by the National Heart, Lung and Blood Institute, as well as by the Institutional Review Board of each participating institution. Total study participation will last about one year.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 16 years old
* Physician-diagnosed asthma for at least one year
* At least one severe asthma exacerbation in the previous year
* Use of asthma medications (daily controller medication [ICS or leukotriene inhibitor] or inhaled β2-agonist [at least three days per week]) for at least six months in the previous year
* Vitamin D insufficiency (i.e., serum vitamin D (25(OH)D level <30 ng/ml (75 nmol/L))
* FEV1 ≥70 % of predicted
* Positive bronchodilator response (i.e., increase in FEV1 ≥8% from baseline after inhaled short acting beta agonist or increased airway responsiveness to methacholine (PC20 ≤8 mg/ml if not on ICS or PC20 ≤16 mg/ml if on ICS)
* Study protocol (i.e., age-appropriate dose of Fluticasone and no other asthma controller medications) approved by the child's regular doctor
* Parental consent and child's assent to participate in the study.

Additional inclusion criteria applied after the run-in period, to be eligible for randomization:

* Adherence with ICS and study medication (≥75% use [at least 21 of 28 days]) during the run-in period
* Willingness to be randomized and complete study

Exclusion Criteria:

* Serum calcium >10.8 mg/dl
* Serum 25(OH) D <14 ng/ml (35 nmol/L)
* Chronic respiratory disorder other than asthma
* Severe asthma (intubation for asthma at any time OR ≥3 hospitalizations for asthma in previous year OR ≥6 severe asthma exacerbations in previous year)
* Hepatic/renal disease, rickets, malabsorption, or other diseases that would affect vitamin D metabolism
* Current smoking, or former smoking if ≥5 pack-years
* Immune deficiency, cleft palate or Down's syndrome
* Treatment with anticonvulsants or ≥1,000 IU/day of vitamin D2 or D3
* Chronic oral corticosteroid therapy
* Inability to perform acceptable spirometry
* Use of investigational therapies or participation in trials 30 days before or during the study
* Participant is currently breast feeding an infant
* Pregnancy
* Weight less than 10 kg
* Plans to move out of the study site area in the next year

Additional exclusion criteria applied after the run-in period:

* Any severe asthma exacerbation during the run-in period
* Need for asthma medications other than ICS and p.r.n. rescue inhalers during the run-in period

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Celedón, MD, DrPH, Principal Investigator — University of Pittsburgh; Stephen Wisniewski, PhD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - University of California - San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han YY, Forno E, Bacharier LB, Phipatanakul W, Guilbert TW, Cabana MD, Ross K, Blatter J, Rosser FJ, Durrani S, Luther J, Wisniewski SR, Celedon JC. Vitamin D supplementation, lung function and asthma control in children with asthma and low vitamin D levels. Eur Respir J. 2021 Oct 28;58(4):2100989. doi: 10.1183/13993003.00989-2021. Print 2021 Oct. PMID 34326185
- [Derived] Forno E, Bacharier LB, Phipatanakul W, Guilbert TW, Cabana MD, Ross K, Covar R, Gern JE, Rosser FJ, Blatter J, Durrani S, Han YY, Wisniewski SR, Celedon JC. Effect of Vitamin D3 Supplementation on Severe Asthma Exacerbations in Children With Asthma and Low Vitamin D Levels: The VDKA Randomized Clinical Trial. JAMA. 2020 Aug 25;324(8):752-760. doi: 10.1001/jama.2020.12384. PMID 32840597

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 595 participants assessed for eligibility, 192 finished run-in and were randomized.
Period: Overall Study
Arm/Group | Vitamin D3 | Placebo
Started | 96 | 96
Completed | 92 | 88
Not Completed | 4 | 8
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 96 | 96 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.5) | 9.7 (2.5) | 9.8 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 33 | 77
  Male | 52 | 63 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 89 | 90 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race abd ethnicity were ascertained per parental report. "Other race" includes American Indian, Alaskan Native, mixed, and other reported as "other".
  Participants
    Race: White | 27 | 32 | 59
    Race: Black | 51 | 49 | 100
    Race: Other Race | 18 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 96 | 96 | 192
Parental Education [Count of Participants; unit: Participants] — Population: 2 participants from the Vitamin D3 group and 1 participant from the placebo group did not have information on parental education
  Participants
    number analyzed (Participants) | 94 | 95 | 189
    High school or less | 21 | 20 | 41
    Some college | 22 | 22 | 44
    Completed college | 37 | 32 | 69
    Postgraduate education | 14 | 21 | 35
Household smoke exposure before age 2 years [Count of Participants; unit: Participants] — Population: 2 participants from Vitamin D3 group and 2 participants from Placebo gorup did not have information on household smoke expousre before age 2 years
  Participants
    number analyzed (Participants) | 94 | 94 | 188
    (all) | 31 | 32 | 63
Current household smoke exposure [Count of Participants; unit: Participants] — Population: 3 participants from Vitamin D3 group and 3 participants from Placebo group did not have information on household smoke exposure during the study
  Participants
    number analyzed (Participants) | 93 | 93 | 186
    (all) | 25 | 22 | 47
Season of enrollment [Count of Participants; unit: Participants]
  January-March | 30 | 25 | 55
  April-June | 26 | 26 | 52
  July-September | 22 | 22 | 44
  October-December | 18 | 23 | 41
Asthma Control Test score >19 [Count of Participants; unit: Participants] — The Asthma Control Test (ACT) was administered to participants aged 12 years or older, and the Childhood Asthma Control Test (C-ACT) was administered to participants aged 6 to 11 years. The ACT is calculated based on 5 self-administered questions and has a score ranges of 5 to 25. The C-ACT is calculated based on 7 questions (3 answered by the parent and 4 answered with the child's input) and has a score range of 0 to 27. For both, a higher score indicates better symptom control, and a score greater than 19 indicates well-controlled asthma symptoms.
  Participants | 76 | 73 | 149
Body Mass Index z-score [Mean (Standard Deviation); unit: z-score] — A body mass index z-score is a measure of relative weight adjusted for the child's age and sex. BMI z-scores were calculated using US Centers for Disease Control and Prevention (CDC) equations that create z-scores and percentiles for a child's sex and age. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher weight. Population: 1 participant in the Vitamin D3 group did not have a valid BMI z-score
  z-score
    number analyzed (Participants) | 95 | 96 | 191
    (all) | 0.9 (1.1) | 0.9 (1.3) | 0.9 (1.2)
No. of severe exacerbations in the previous year [Median (Inter-Quartile Range); unit: exacerbations] — A severe asthma exacerbation was defined as the occurrence of either (1) use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or (2) a hospitalization or ED visit because of asthma, requiring systemic corticosteroids Population: 8 participants in the Vitamin D3 group and 10 participants in the placebo group did not have such information
  exacerbations
    number analyzed (Participants) | 88 | 86 | 174
    (all) | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Vitamin D [Mean (Standard Deviation); unit: ng/mL] | 22.5 (4.6) | 22.8 (4.6) | 22.6 (4.6)
FEV1 [Mean (Standard Deviation); unit: % predicted] — Forced Expiratory Volume in the first second (FEV1) refers to the maximum amount of air that the subject can forcibly expel during the first-second following maximal inhalation. All participants performed spirometry following American Thoracic Society/European Respiratory Society guidelines. Calculated using reference values from the third National Health and Nutrition Examination Survey. Values 80% of predicted or greater are considered normal.
  % predicted | 93.9 (15.8) | 90.6 (17.3) | 92.2 (16.6)
FEV1/FVC [Mean (Standard Deviation); unit: % predicted] — FEV1/FVC is the ratio of the forced expiratory volume in the first one second (FEV1) to the forced vital capacity (FVC, the total amount of air exhaled) of the lungs. A reduced FEV1/FVC represents obstruction of airflow. All participants performed spirometry following American Thoracic Society/European Respiratory Society guidelines. Calculated using reference values from the third National Health and Nutrition Examination Survey. Values 80% of predicted or greater are considered normal.
  % predicted | 91.5 (9.3) | 89.6 (10.1) | 90.6 (9.7)
Asthma Control Test score [Mean (Standard Deviation); unit: units on a scale] — For participants aged ≥12 years, asthma control was assessed using the Asthma Control Test (ACT [score range, 5-25].
  For participants aged <12 (6-11) years, asthma control was assessed using Childhood ACT (C-ACT [score range,0-27].
  For both tests, higher scores mean better symptom control, and more than 19 points is considered well controlled asthma.
  units on a scale | 22.0 (3.2) | 21.3 (3.6) | 21.7 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Days to a Severe Asthma Exacerbation
Description: A severe asthma exacerbation is defined as an exacerbation that meets either of these criteria: 1) Use of systemic corticosteroids (tablets, suspension, or injection), or an increase from a stable maintenance dose, for at least 3 days OR 2) A hospitalization or ER visit because of asthma, requiring systemic corticosteroids.
Time Frame: 48 weeks
Population: Intent to treat population across the 48-week study period
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 96 | 96
Days | 240 (105.8) | 253 (101.3)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.63, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.69 to 1.85]

2. Secondary Outcome: Days to Viral-induced Severe Exacerbation
Description: A severe viral asthma exacerbation is defined as a severe asthma exacerbation [defined as an exacerbation that meets either of these criteria: 1) Use of systemic corticosteroids (tablets, suspension, or injection), or an increase from a stable maintenance dose, for at least 3 days OR 2) A hospitalization or ER visit because of asthma, requiring systemic corticosteroids] along with a positive respiratory viral panel from a nasal blow collected within 72 hours of the exacerbation.
Time Frame: 48 weeks
Population: In Vitamin D3 gorup, 82 with time to viral exacerbation were included in the analysis (14 first exacerbations not tested). In Placebo group, 83 with time to viral exacerbation were included in the analysis (13 first exacerbations not tested)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 82 | 83
Days | 272 (87.8) | 281 (83.6)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.46, Regression, Cox; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.63 to 2.75]

3. Secondary Outcome: Proportion of Participants in Whom Fluticasone Dose Was Halved at Visit 6
Description: In the absence of moderate or severe asthma exacerbations, participants may have their dose of inhaled corticosteroids (ICS) reduced by 50% if the following criteria are met at visit 6 (halfway through the Trial Phase):
  * Asthma Control Test (ACT) score greater than 19
  * Both pre-bronchodilator FEV1 and FEV1/FVC ≥80% of predicted
  * Use of ≤4 puffs of a rescue inhaler per week
  * ≤1 day per month with asthma symptoms preventing full participation in usual daily activities
  * Clinician's judgment regarding adequate asthma control
Time Frame: 24 weeks
Population: In the Vitamin D3 group, 91 subjects with data on reduction in the dose of inhaled corticosteroids (4 withdrew before 24 wk, 1 missed 24-wk visit). In the Placebo group, 91 subjects had data on reduction in the dose of inhaled corticosteroids (4 withdrew before 24 wk, 1 missed 24-wk visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 28 | 29
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.66 to 1.52]

4. Secondary Outcome: Average Cumulative Prescribed Dose of ICS at the End of the Trial
Description: The average cumulative dose of inhaled corticosteroids (ICS) during the study period
Time Frame: 48 weeks
Population: Intent to treat population across the 48-week study period
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 96 | 96
mg | 59.6 (22.9) | 55.2 (14.5)
Statistical Analysis 1: Comparison: Vitamin D3 vs Placebo; Test type: Superiority; p = 0.049, Regression, Linear; Mean Difference (Final Values) = 4.40, 95% CI 2-sided [0.001 to 8.80]

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: A hospitalization for an asthma exacerbation was considered a serious adverse event.
Arm/Group | Vitamin D3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 9/96 | 7/96
Other Adverse Events (participants affected / at risk) | 5/96 | 4/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 (N=96) | Placebo (N=96)
Hospitalization for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (6)
eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
severe neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia/otitis/hives (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 (N=96) | Placebo (N=96)
Fractures (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) — Fractures

LIMITATIONS AND CAVEATS:
Limited statistical power to determine if vitamin D supplementation prolongs the time to a severe asthma exacerbation in children with vitamin D level <20 ng/ml.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT02687815/Prot_SAP_000.pdf